CLINICAL TRIAL: NCT04587401
Title: The Effects of Anesthesia on Cerebral Perfusion Identified by Transcranial Doppler During Lumbar Surgery in Prone Position in Patients With High Blood Pressure.
Brief Title: The Effects of Anesthesia on Cerebral Perfusion in Patients With High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, yesim cetintas, Principal investigator, Akdeniz University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AkdenizU-438
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2020-09

CONDITIONS: Lumbar Disc Disease; Lumbar Spinal Stenosis; Lumbar Disc Herniation; Lumbar Fracture
Keywords: transcranial doppler ultrasonography; high blood pressure; cerebral perfusion; prone position
MeSH Terms: conditions — Intervertebral disc disease; Spinal Stenosis; Intervertebral Disc Displacement; Fractures, Bone; Hypertension

STUDY DESIGN:
Intervention Model Description: Patients, aged between 18 and 85, who were scheduled for lumbar surgery under general anesthesia by neurosurgery department and were classified as Class I, II, and III according to the ASA (American Association of Anesthesiologists) classification, were included in the study.
Who Masked: Participant, Care Provider
Masking Description: Patients with mental retardation, with brain tumor, head trauma, cerebral aneurysm, cerebrovascular accident, dementia, psychiatric disease, and carotid stenosis were excluded from the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normotensive patients (Experimental): Cerebral perfusion of normotensive patients who will have lumbar surgery at the prone position will be measured by transcranial doppler ultrasonography
  Interventions: Procedure: normotensive patients
- patients with high blood pressure diagnosis (Experimental): Cerebral perfusion of patients with high blood pressure diagnosis who will have lumbar surgery at the prone position will be measured by transcranial doppler ultrasonography
  Interventions: Procedure: patients with hypertension diagnosis
- patients who do not know they are hypertensive but actual blood pressure is high (Experimental): cerebral perfusion of patients who do not have high blood pressure diagnosis but actual preoperative blood pressure is higher than normal levels will be measured by transcranial doppler ultrasonography during lumbar surgery
  Interventions: Procedure: patients who do not know they are hypertensive but actual blood pressure is high

INTERVENTIONS:
Procedure: normotensive patients — patients who do not have high blood pressure diagnosis and actual blood pressure is within the normal range
  Arms: normotensive patients
Procedure: patients with hypertension diagnosis — Patients who have high blood pressure diagnosis
  Arms: patients with high blood pressure diagnosis
Procedure: patients who do not know they are hypertensive but actual blood pressure is high — patients with preoperative high blood pressure, who do not know they are hypertensive
  Arms: patients who do not know they are hypertensive but actual blood pressure is high

SUMMARY:
High blood pressure is a serious and common health problem. This disease affects 1 billion people all over the world and responsible for 7,1 million deaths. Trials involving more than 1 million people state that stroke incidence rises as blood pressure rises. The effects of high blood pressure on cerebral perfusion is not well realized. Intraoperative blood pressure management of patients with high blood pressure is not well known. And it is still not clear how autoregulation of cerebral perfusion is affected by high blood pressure.

Systemic arterial pressure changes have little effect on cerebral perfusion. This is regulated by changes of precapillary resistance. When systemic arterial blood pressure drops, it is regulated by vasodilatation of arteriolar smooth muscles. And when systemic blood pressure rises, it is regulated by vasoconstriction of arterioles. Cerebral perfusion is well preserved between 50-125 mmHg changes of mean arterial blood pressure (MAP). Patients with high blood pressure have higher ranges. Patients with chronic high blood pressure can better tolerate higher blood pressures. But even physiologic drops of systemic blood pressure can cause ischemia.

Anesthetic drugs have variable effects on cerebral blood flow and physiology. The drugs used with anesthetic drugs, the noxious stimulus of surgery, intracranial compliance, blood pressure, and carbon dioxide pressure can all alter and complicate these effects. Anesthetic drugs must be selected carefully in patients with high blood pressure. It is still investigated whether, management of blood pressure under anesthesia, should be individualized.

For patients with high blood pressure, some neuromonitorization technics have been evaluated to prevent neurologic complications under anesthesia. But there is not a technic, which is considered as a gold standard. Cerebral blood pressure has been studied by, nitrous oxide method, krypton uptake method, and xenon injection methods previously. Near-infrared spectroscopy (NIRS) is the best monitorization technic of intracranial pressure (ICP), cerebral blood flow (CBF), and cerebral metabolism. But it can not be applied to all patients. Recently, it is possible to measure blood flow of cerebrum with transcranial Doppler ultrasound in anesthesia practice.

In this trial, the investigators aim to evaluate cerebral perfusion of hypertensive patients with transcranial Doppler during lumbar disc surgery to optimize the blood pressure under anesthesia.

To best of our knowledge, there is no trial evaluating cerebral perfusion of hypertensive patients with transcranial Doppler ultrasound.

DETAILED DESCRIPTION:
In this trial, the investigators aim to evaluate the cerebral perfusion of patients with transcranial doppler ultrasound (TCD) and near-infrared spectroscopy (NIRS) during lumbar disc surgery.

The investigators will divide participants into three groups according to their blood pressure history after preoperative evaluation of the participants.

The investigators will enroll normotensive participants in group 1(control group). Participants with diagnosis of high blood pressure will be enrolled to group 2. In the third group, participants who don't have any diagnosis of high blood pressure, but actual blood pressure is higher than the physiological levels at the preoperative evaluation will be enrolled to group 3.

First measurements of TCD and NIRS, will be performed at preoperative period. Second measurements will be obtained after anesthesia induction. Third measurement will be performed after prone position. Forth measurement will be taken after 1 hour of surgical incision. The last measurement will be performed at the postoperative period.

During all these measurements, blood gas samples, invasive arterial blood pressures, pulse variation index (PVI), electrocardiography (ECG), peripheral oxygen saturation (SpO2), peak pressure of airway and end-tidal carbon dioxide (EtCO2) levels will also be recorded.

All participants will be evaluated for their cognitive functions with mini-mental and confusion assessment method (cam) tests at the preoperative and postoperative periods.

ELIGIBILITY:
Inclusion Criteria: Clinical diagnosis of lumbar stenosis Clinical diagnosis of lumbar fracture Clinical diagnosis of lumbar mass -

Exclusion Criteria: Patients who had an intracranial incident Patients with anesthetic risk classification higher than American Society of Anesthesiology (ASA) 3 Carotid atherosclerosis

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Mean cerebral perfusion pressure of hypertensive patients under anesthesia | time from the preoperative period of the surgery until the postoperative 24th hour of the surgery
  Mean cerebral perfusion pressure will be measured by transcranial doppler ultrasonography under anesthesia

SECONDARY OUTCOMES:
Comparison of transcranial doppler and near-infrared spectroscopy for determining of cerebral perfusion | time from the preoperative period of the surgery until the postoperative 24th hour of the surgery
  Transcranial doppler and near-infrared spectroscopy measurements will be compared by neurocognitive tests after the surgery

OTHER OUTCOMES:
Determination of changes of the cerebral perfusion in patients with actual high blood pressure who has not been diagnosed for hypertension before. | time from the preoperative period of the surgery until the postoperative 24th hour of the surgery
  Mean cerebral arterial pressure of patients with actual high blood pressure but without hypertension diagnosis will be measured by transcranial doppler ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Neval Boztug, Prof, Study Director — Akdeniz University Medical School Anesthesiology and Reanimation Department
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No